CLINICAL TRIAL: NCT00907075
Title: Pilot Study to Assess Adherence to a Novel Eating System in Men and Women With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: Provident Clinical Research (Other)
Responsible Party: Richard Black, PhD/VP, Nutrition, Kraft Foods
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRV-08012; PRV-08012V1.9
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; nutrition; diet; foods
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NES With Energy Restriction (Active Comparator)
  Interventions: Behavioral: NES With Energy Restriction
- NES Without Energy Restriction (Active Comparator)
  Interventions: Behavioral: NES Without Energy Restriction

INTERVENTIONS:
Behavioral: NES With Energy Restriction — The NES will be administered based upon the individual's calculated daily energy requirement, with an energy deficit of approximately 500 kilocalories.
  Arms: NES With Energy Restriction
Behavioral: NES Without Energy Restriction — The NES will be administered based upon the individual's calculated daily energy requirement.
  Arms: NES Without Energy Restriction

SUMMARY:
The purpose of this pilot study is to assess adherence to a Novel Eating System (NES) with and without energy restriction.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-79 years of age, inclusive.
2. Diagnosis of type 2 diabetes, at least nine months prior to screening.
3. Stable use of oral hypoglycemic medication for at least two months prior to screening.
4. Body mass index (BMI) ≥25.0 and <45.0 kg/m2 at screening.
5. Willingness to follow a novel eating plan, which may be energy restricted to promote weight loss, throughout the trial.

Exclusion Criteria:

1. History or diagnosis of type 1 diabetes mellitus.
2. Poorly controlled type 2 diabetes mellitus (HbA1C ≥9.0%).
3. Weight loss or gain >10 lb (4.5 kg) in the two months prior to screening.
4. Abnormal laboratory test results of clinical importance.
5. History of gastrointestinal surgery for weight-reducing purposes.
6. Poorly controlled hypertension.
7. A clinically important medical or other condition.
8. Any major trauma or major surgical event within three months of screening.
9. Use of injected medications for glucose control within four weeks prior to screening.
10. Use of weight loss medications, supplements, programs, or meal replacement products within two months of screening.
11. Unstable use of foods, dietary supplements, herbals or medications, other than allowed medications, that have the potential to influence carbohydrate or lipid metabolism.
12. Pregnancy
13. Any history of extreme eating habits or an eating disorder diagnosed by a health professional.
14. Recent history of (within 12 months of visit 1) or strong potential for alcohol or substance abuse.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Average percent deviations from the assigned eating system score for full days, meals, and snacks for each group during each evaluation period throughout the intervention (days 23-28 and days 51-56). | 10 weeks

SECONDARY OUTCOMES:
Change in 24 hour mean circulating glucose level from baseline to end of treatment. | 10 weeks
Change in fasting plasma glucose and insulin from baseline to end of treatment. | 10 weeks
Change in lipid parameters (Total cholesterol, LDL-C, HDL-C, triglycerides) from baseline to end of treatment. | 10 weeks
Change in dietary macronutrient composition from baseline to end of treatment. | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Maki, PhD, Study Director — Provident Clinical Research & Consulting, Inc.
Locations (2):
- United States (2):
  - Provident Clinical Research & Consulting, Inc., Addison, Illinois
  - Provident Clinical Research & Consulting, Inc., Bloomington, Indiana